CLINICAL TRIAL: NCT02401100
Title: Anastomotic Leakage After Anterior Resection for Rectal Cancer - Predictive Biomarkers and Rectal Blood Flow
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: UmU-AL-01
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2018-10

CONDITIONS: Anastomotic Leak
Keywords: Rectal Neoplasms
MeSH Terms: conditions — Anastomotic Leak; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Preoperative and postoperative blood samples. Postoperative drain fluid samples. Tissue samples from the perianastomotic region taken perioperatively.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether reduced rectal blood flow is associated with the extent of surgery when performing an operation to remove rectal cancer. The investigators also aim to describe any relation of reduced rectal blood flow, as well as raised inflammatory biomarkers in blood and tissue, to the occurrence of anastomotic leakage. The patients will be recruited at Umeå University Hospital and all patients who are planned to undergo anterior resection for rectal cancer and able to consent are eligible for this study. Rectal blood flow measurements will be conducted with Laser-Doppler technology using noninvasive measuring probes. Preoperative and postoperative blood sampling as well as postoperative drain fluid collection will take place. Perianastomotic tissue will also be collected. In the postoperative period, any occurrence of surgical complications especially anastomotic leakage, will be noted. Blood flow and biomarkers will be assessed in relation to type of mesorectal excision (total or partial) and correlated to anastomotic leakage. Standard statistical tools will be utilized, such as parametric, non-parametric tests and logistic regression, as appropriate. The study will recruit approximately 40 patients during three consecutive years.

ELIGIBILITY:
Inclusion Criteria:

* Planned anterior resection for rectal cancer
* Willing to participate

Exclusion Criteria:

* Not willing to participate
* Unable to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rectal cancer who undergo anterior resection for rectal cancer at Umeå University Hospital.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Blood flow measurements | Start and end of operation
  Laser-Doppler blood flow measurements of the rectal mucosa perfusion below and distal to the anastomosis.

SECONDARY OUTCOMES:
Anastomotic leakage | 90 days postoperatively
  The occurrence of anastomotic leakage, as defined by the International Study Group for Rectal Cancer (ISREC).

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rutegård, M.D., Ph.D., Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Back E, Brannstrom F, Svensson J, Rutegard J, Matthiessen P, Haapamaki MM, Rutegard M. Mucosal blood flow in the remaining rectal stump is more affected by total than partial mesorectal excision in patients undergoing anterior resection: a key to understanding differing rates of anastomotic leakage? Langenbecks Arch Surg. 2021 Sep;406(6):1971-1977. doi: 10.1007/s00423-021-02182-0. Epub 2021 May 18. PMID 34008097